CLINICAL TRIAL: NCT07179419
Title: Evaluation of the Long-term Therapeutic Effect of High-Intensity Focused Ultrasound (HIFU) Treatment in Patients With Rectal Endometriosis
Acronym: ENDO HIFU FU
Status: Recruiting | Type: Observational
Sponsor: EDAP TMS S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: HIFU/F/21.04
Record Dates: First submitted 2025-09-11; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Endometriosis
Keywords: HIFU; FocalOne; Rectal Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate the long-term effects of HIFU treatment for rectal endometriosis.

DETAILED DESCRIPTION:
This study evaluates the long-term effects of HIFU treatment on endometriosis symptoms in patients who have received this treatment. The patients included will have participated in the following studies: HIFU/F/13.12, ENDO HIFU R1, and ENDO HIFU R2.

Patients will complete an electronic questionnaire and receive a telephone call to monitor these parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been treated with HIFU for rectal endometriosis included in study HIFU/F/13.12, study HIFU/F/20.01 (ENDO HIFU R1) or study HIFU/F/21.12 (ENDO HIFU R2)
* Agreeing to participate in the study
* Patients with internet access so that they can complete the questionnaires electronically.

Exclusion Criteria:

* Patients deprived of their liberty following a judicial or administrative decision,
* Patients under guardianship or conservatorship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who received HIFU treatment for rectal endometriosis as part of studies HIFU/F/13.12, HIFU/F/20.01, and HIFU/F/21.12.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Compare the SF36 score assessed before HIFU treatment with that assessed in the long term after HIFU treatment. | every year during 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital de la Croix Rousse, Lyon, France